CLINICAL TRIAL: NCT03721744
Title: A Phase II/III Randomized, Open-Label Clinical Study of GB201 in Combination With Weekly Paclitaxel and Low-dose Gemcitabine in Patients With Metastatic Pancreatic Cancer Following Chemotherapy Failure
Brief Title: A Study of GB201 in Combination With Weekly Paclitaxel and Low-dose Gemcitabine in Patients With Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: 1Globe Health Institute LLC (Industry)
Responsible Party: Sponsor
Organization: 1Globe Biomedical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STEMNESS-PANC
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GB201+Paclitaxel+Gemcitabine (Experimental): Patients randomized to Arm 1 will receive GB201 in combination with weekly paclitaxel and low-dose gemcitabine, with one treatment cycle defined as 4 weeks (28 days). GB201 will be administered orally, twice daily, with doses separated by approximately 8-12 hours. GB201 administration will begin 2-5 days prior to the first infusion of paclitaxel and low-dose gemcitabine.
  Paclitaxel and low-dose gemcitabine will be administered on Days 1, 8 and 15 of every 28-day cycle.
  Interventions: Drug: GB201; Drug: Paclitaxel; Drug: Gemcitabine
- Standard of care treatment options (Active Comparator): Patients randomized to Arm 2 will receive one of the standard of care treatment options assigned by the Investigator for each patient prior to starting protocol treatment, including gemcitabine, capecitabine, 5-FU/LV, Onivyde plus 5- FU/LV (if Onivyde is available in the country/region) or best supportive care (BSC). Patients who have failed gemcitabine previously and were randomized to Arm 2 will not be eligible to receive gemcitabine as a treatment option.
  Interventions: Other: Standard of care treatment options

INTERVENTIONS:
Drug: GB201 — GB201 will be administered orally, twice daily, with doses separated by approximately 8-12 hours. GB201 administration will begin 2-5 days prior to the first infusion of paclitaxel and low-dose gemcitabine
  Arms: GB201+Paclitaxel+Gemcitabine
Drug: Paclitaxel — Paclitaxel 80 mg/m^2 will be administered intravenously starting on Day 1 of Cycle 1. This regimen will be repeated on Days 1, 8 and 15 of every 28-day cycle
  Arms: GB201+Paclitaxel+Gemcitabine
Drug: Gemcitabine — Low-dose gemcitabine 600 mg/m^2 will be administered intravenously following completion of paclitaxel infusion. This regimen will be repeated on Days 1, 8 and 15 of every 28-day cycle.
  Arms: GB201+Paclitaxel+Gemcitabine
Other: Standard of care treatment options — Patients will receive one of the standard of care treatment options assigned by the Investigator for each patient prior to starting protocol treatment, including Gemcitabine, capecitabine, 5-FU/LV, Onivyde plus 5-FU/LV (if Onivyde is available in the country/region) or best supportive care (BSC).
  Other Names: BSC
  Arms: Standard of care treatment options

SUMMARY:
This is a Phase II/III Randomized, Open-Label Clinical Study of GB201 in Combination with Weekly Paclitaxel and Low-dose Gemcitabine in Patients With Metastatic Pancreatic Cancer Following Chemotherapy Failure

ELIGIBILITY:
INCLUSION CRITERIA

1. Written, signed consent for trial participation in accordance with applicable ICH guidelines.
2. Must have histologically or cytologically confirmed advanced pancreatic adenocarcinoma that is metastatic.
3. Patients who are candidates for and have access to gemcitabine-nab-paclitaxel or are candidates for FOLFIRINOX/mFOLFIRINOX must have received these standard of care regimens before randomization.
4. Must have one or more evaluable metastatic tumors by RECIST 1.1.
5. Must have ECOG Performance Status of 0 or 1.
6. Must have life-expectancy of > 12 weeks.
7. Must be ≥ 18 years of age.
8. For male or female patients of child producing potential: must agree to use contraception or take measures to avoid pregnancy.
9. Adequate biological parameters：

   * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L
   * Platelet count ≥ 100,000/mm^3 (100 × 10^9/L).
   * Hemoglobin (Hgb) ≥ 9 g/dL.
   * AST (SGOT) and ALT (SGPT) ≤ 2.5 × institutional upper limit of normal (ULN) [5 ×ULN in presence of liver metastases]
   * Total bilirubin ≤ 1.5 × institutional ULN. If total bilirubin is > ULN, it must be non-rising for at least 3 days.
   * Serum creatinine within normal limits or calculated clearance > 60 mL/min/1.73 m^2.
10. Acceptable coagulation studies.
11. No clinically significant abnormalities on urinalysis.
12. Patient must have adequate nutritional status.
13. Pain symptoms should be stable (of tolerable Grade 2 or less).
14. Only patients with available archival tumor tissue must consent to submit block of tumor tissue.
15. The patient is not receiving therapy in a concurrent clinical study.

EXCLUSION CRITERIA

1. Anti-cancer chemotherapy, radiotherapy, biologic therapy or immunotherapy administered two weeks prior to the first planned dose of study medication. Investigational agents administered within four weeks of first planned dose of study medication.
2. Patients with any unresolved lingering toxicity > Grade 2 from prior treatment will be excluded.
3. Patient who were intolerant to prior taxane treatment.
4. Major surgery within 4 weeks prior to randomization.
5. Patients with any known brain or leptomeningeal metastases are excluded, even if treated.
6. Patients with clinically significant pleural effusion or ascites.
7. Patient with gastrointestinal disorder(s) which could significantly impede the absorption of an oral agent.
8. Prior treatment with napabucasin or participation in a clinical trial evaluating napabucasin.
9. Uncontrolled inter-current illness.
10. Known hypersensitivity to gemcitabine, taxanes or any of their excipients.
11. Uncontrolled chronic diarrhea ≥ grade 2 at baseline.
12. Patients being treated with any coumarins.
13. Patients with a history of other malignancies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2018-10-25 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 30 months
  The primary objective of this study is to compare overall survival (OS) of patients with metastatic pancreatic adenocarcinoma treated with GB201 in combination with weekly paclitaxel and Low-dose gemcitabine versus standard of care treatment options.

SECONDARY OUTCOMES:
Progression free survival (PFS) | 30 months
  Defined as the time from randomization to the first objective documentation of disease progression or death due to any cause.
Objective response rate (ORR) | 30 months
  Defined as the proportion of patients with a documented complete response or partial response (CR + PR) based on RECIST 1.1
Disease control rate (DCR) | 30 months
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1
Quality of Life (QoL) | 30 months
  European Organization for Research and Treatment of Cancer Quality of Life questionnaire（EORTC-QLQ-C30), is a self-administered cancer specific questionnaire with multi-dimensional scales. It consists of both multi-item scales and single item measures, including five functional domains, a global quality of life domain, three symptom domains, and six single items. For each domain or single item measure a linear transformation will be applied to standardize the raw score to range between 0 and 100. The endpoints in QoL analysis are the mean EORTC QLQ-C30 QoL change scores from baseline for the physical function and global health status/quality of life subscale scores. After transformation, higher scores in these two subscales mean better outcome
Safety by reporting the adverse events and serious adverse events | 30 months
  Assessment of safety of GB201 by reporting of adverse events and serious adverse events.

CONTACTS AND LOCATIONS:
Locations (38):
- China (32):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijng Cancer Hospital, Beijing, Beijing Municipality
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - SUN YAT-SEN University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - People's Hospital of Hunan Province, Changsha, Hunan
  - The Third Xianya Hospital of Central South University, Changsha, Hunan
  - The 81 Hospital of the Chinese People Liberation Army, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - The First Bethune Hospital of Jilin University, Changchun, Jilin
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - East Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute Hospital, Tianjin, Tianjin Municipality
  - Sir Run Shaw Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang
  - The First Affiliated Hospital Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Hospital of Jiaxing, Jiaxing, Zhejiang
- France (3):
  - Institut de Cancerologie de Lorraine, Bourgogne
  - Unité de Recherche Clinique en Cancérologie, Institut de cancérologie et d'hématologie, Brest
  - Centre Antoine Lacassagne, Nice
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario HMN Sanchinarro, Madrid
  - Hospital Universitario La Paz, Madrid